CLINICAL TRIAL: NCT02865642
Title: CISS: Cortical Ischemic Stroke and Serotonin - Effects of Serotonergic Neuromodulation on Behavioural Recovery and Motor Network Plasticity After Cortical Ischemic Stroke: a Longitudinal, Placebo-controlled Study
Brief Title: Cortical Ischemic Stroke and Serotonin
Acronym: CISS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 3070; 2016-00417 (Other: KEK)
Record Dates: First submitted 2016-08-04; First posted 2016-08-12 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Stroke
Keywords: Stroke; Serotonin; Hand Paresis
MeSH Terms: conditions — Stroke | interventions — Selective Serotonin Reuptake Inhibitors; Escitalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Serotonin Uptake Inhibitors (Experimental): Treatment 1: Starting with Escitalopram 5mg/day at the baseline-visit (day 14 (+-7) post stroke) for 7 days followed by a weekly dosage increase of 5mg/day till target dose of Escitalopram 20mg/day.
  Subjects will remain on Escitalopram 20mg/day until visit 3 (day 90 (+-14) post stroke) followed by dosage reduction of Escitalopram 10mg/day for one week.
  Interventions: Drug: Serotonin Uptake Inhibitors
- Placebo (Placebo Comparator): Treatment 2: Starting with Placebo 5mg/day at the baseline-visit (day 14 (+-7) post stroke) for 7 days followed by a weekly dosage of 5mg/day till target dose of Placebo 20mg/day.
  Subjects will remain on Placebo 20mg/day until visit 3 (day 90 (+-14) post stroke) followed by Placebo 10mg/day for one week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Serotonin Uptake Inhibitors
  Other Names: Escitalopram, Cipralex
  Arms: Serotonin Uptake Inhibitors
Drug: Placebo
  Arms: Placebo

SUMMARY:
In this study the investigators want to test the hypotheses that, serotonergic neuromodulation increases perilesional neuroplasticity, leading to improved behavioural outcomes through a more efficient allocation of functional resources, greater structural reorganization and less remapping via alternative circuits.

DETAILED DESCRIPTION:
Neuroplasticity, i.e. the human brain's innate capacity to structurally remodel and functionally reorganize its neural networks, is essential for recovery of impaired sensorimotor function after focal ischemic injury. However, the potential for spontaneous recovery in the adult brain is limited and needs to be augmented through rehabilitative programs, e.g. intensive exercise, brain stimulation or pharmacologic neuromodulation.

Clinical studies have shown that post-stroke recovery can be augmented by long-term administration of selective serotonin reuptake inhibitors (SSRI). Serotonin modulates excitatory glutamatergic neurotransmission and induces long-term potentiation (LTP), an important mediator of neuroplasticity that supports sensorimotor learning in the healthy brain and reorganization in the post-stroke perilesional cortex. Preliminary data indicate that a single dose of the SSRI Escitalopram is sufficient to induce LTP-like effects in the motor cortex of healthy volunteers (measured by repetitive transcranial magnetic stimulation (rTMS)), and to increase the efficiency of large-scale functional connectivity networks engaged in tactile object manipulation ( measured with functional magnetic resonance imaging (fMRI)).

The investigators thus hypothesize that serotonergic neuromodulation might enhance post-stroke recovery through enlarged plasticity and processing efficiency along integrated neuronal networks, leading to reinforced connectivity and behavioural performance.

To test this hypothesis, the investigators aim to conduct a longitudinal, double blind, placebo-controlled trial in two neurological centers. The investigators aim to test the effect of a daily-administered single dose of Escitalopram over a three months period after cortical ischemic stroke to promote plasticity changes in the perilesional zone of primary sensorimotor cortices (S1 and M1). The investigators will apply behavioural measures of hand function, rTMS and advanced magnetic resonance (MR) imaging techniques as outcome variables.

The investigators will measure hand function kinematics with a data glove to better understand the contribution of effort to hand function recovery and brain activation. Moreover, the investigators intend to apply MR-Spectroscopy of the perilesional premotor cortex, guided by real-time fMRI analysis, as a tool to assess local glutamatergic transmission. Measurements of plasma drug levels and determination of genetic polymorphisms of the Escitalopram-metabolizing genes will help them to assess and control for interindividual variance in Escitalopram bioavailability.

The investigators expect that SSRI-augmented neuroplasticity will lead to increased efficiency in the allocation of neuronal resources in the post-stroke brain, resulting in more precise and less effortful movements, facilitation of LTP-like phenomena, increased grey matter volume of spared perilesional premotor cortex and possibly higher glutamate peaks in the same areas, as compared to placebo treatment.

By combining standard and innovative methods, this study will provide mechanistic insight into the processes that drive cortical neuroplasticity in the post-stroke human brain. From a clinical perspective, results from the study are expected to provide a scientific rationale to select patients that might benefit from SSRI-augmented neurorehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* First-ever stroke
* Clinically significant contralesional hand plegia or paresis as a main symptom
* Involvement of the pre-and/or postcentral gyri confirmed on diffusion-weighted (DWI) and fluid attenuated inversion recovery (FLAIR) scans.
* Written informed consent

Exclusion Criteria:

* Aphasia or cognitive deficits severe enough to preclude understanding of study purposes
* Prior cerebrovascular events
* Significant stenosis (70-99% according to NASCET) or occlusion of the carotid and intracranial arteries on MR-angiography
* Purely subcortical stroke
* Known brain lesion (tumour, old cerebral haemorrhage)
* Other medical conditions interfering with task performance or SSRI-treatment, specifically: prolonged corrected QT interval (QTc) on electrocardiogram, ongoing drug / alcohol abuse
* Simultaneous intake of medications which can lead to prolonged QTc syndrome known or or suspected hypersensitivity (allergic) to one of the ingredients of Cipralex® or Placebo
* Simultaneous administration of: antidepressants, irreversible non- selective Monoamine Oxidase (MAO) inhibitors, reversible selective MAO inhibitors, reversible non-selective MAO inhibitors, irreversible selective MAO inhibitors, N-methyl-D-aspartate(NMDA)-receptor antagonists/-agonists, dopamine antagonists/-agonists, levodopa, benzodiazepines, amphetamines, methylphenidate, foscarnet, ganciclovir, ritonavir, mianserin, chloroquine, mefloquine, imipenem, penicillin, ampicillin, cephalosporins, metronidazole, isoniazid, levofloxacin, cyclosporin, chlorambucil, vincristine, methotrexate, cytosine arabinoside, lithium, anticholinergics,systemic antihistamines, systemic sympathomimetics
* Conditions interfering with MRI such as patients with magnetic (metallic) particles in the scull or brain, patients with a cardiac pacemaker, deep brain stimulators or cochlear implant.
* Women who are pregnant or breastfeeding
* Women in childbearing age without sufficient birth control (at least 2 contraceptive methods)

Eligibility Criteria for healthy volunteers:

* Normal test-scores at the baseline visit (see section 5.2.2)
* Normal neurological status
* No known brain lesion
* No pregnancy
* Written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-08; Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Effect of escitalopram on sensorimotor network | fMRI at month 9
  To verify higher expression of the sensorimotor network engaged in motor control in the blood oxygenation level dependent (BOLD) response of task-related fMRI (act-fMRI) in patients treated with escitalopram compared to patients treated with placebo after nine months

SECONDARY OUTCOMES:
Imaging patterns of rs-fMRI | rs-fMRI (baseline, month 3, month 9)
  To compare imaging patterns of rs-fMRI and associated behavioral parameters of the verum and placebo group with those of healthy volunteers in the longterm in order to assess the degree of recovery.
Imaging patterns of act-fMRI | act-fMRI, performance of tactile manipulation of objects (baseline, month 3, month 9)
  To compare imaging patterns act-fMRI and associated behavioral parameters of the verum and placebo group with those of healthy volunteers in the longterm from baseline until month 3 and 9 in order to assess the degree of recovery and the associated efficiency in performing tactile manipulation of objects.
Jebsen-Taylor Test (JTT) | JTT, monthly from baseline to month 9
  To calculate the recovery trajectories of subjects post-stroke, relying on motor subtests of the JTT which will be carried out monthly from baseline to month 9.
Mean cortical volume changes | T1 from baseline, month 3, month 9
  To delineate overall mean cortical volume changes in the longterm from baseline until 9 months in high-resolution T1-images to detect structural reorganization post-stroke both perilesional and in distributed large scale networks specifically related to hand motor skill in the verum and placebo group.
Serum concentration of escitalopram | Serum concentration at month 3
  To explore the serum concentration (µg/L) of escitalopram as possibly confounding factors impacting on the study results.
Genetic polymorphisms in genes | Genetic polymorphisms in genes at month 3
  To explore the number of patients with genetic polymorphisms in genes (CYP2P19, ABCB1, CYP3A4 or CYP3A5) as possibly confounding factors impacting on the study results.

OTHER OUTCOMES:
Glutamate/Glutamine concentration | Spectroscopy at baseline, month 3, month 9
  Substudy Center 1: To measure Glutamate/Glutamine concentration post-stroke by MR-Spectroscopy in predefined brain areas (i.e. in the ipsilesional sensorimotor cortex and dorsolateral prefrontal cortex) as possible factor interfering with the recovery process
rTMS | TMS at baseline, month 3, month 9
  Substudy Center 2: To assess for facilitation in the motor system after application of escitalopram, using rTMS in the verum group related to the placebo group.
Number of adverse events due to study medication | Baseline, monthly until month 9
  Number of adverse events due to study medication Safety Endpoint: Experiencing at least one serious adverse event (e.g. death, life-threatening, requires inpatient hospitalization)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Wiest, Principal Investigator — Support Center of Advanced Neuroimaging Institute for Diagnostic and Interventional Neuroradiology Inselspital, University Hospital Bern; Georg Kägi, Principal Investigator — Neurology Department Kantonsspital St. Gallen
Locations (2):
- Switzerland (2):
  - Neurology Department Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Support Center of Advanced Neuroimaging Institute for Diagnostic and Interventional Neuroradiology Inselspital, University Hospital Bern, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krammer W, Missimer JH, Habegger S, Pastore-Wapp M, Wiest R, Weder BJ. Sensing form - finger gaiting as key to tactile object exploration - a data glove analysis of a prototypical daily task. J Neuroeng Rehabil. 2020 Oct 8;17(1):133. doi: 10.1186/s12984-020-00755-6. PMID 33032615